CLINICAL TRIAL: NCT03878758
Title: Comparative User Experiences With BD Nano™ PRO 4mm x 32G Extra Thin Wall Pen Needle vs the Artsana Insupen® Extr3me 4mm x 33G, Artsana Insupen® Extr3me 3.5mm x 34G and the Simple Diagnostics Comfort EZ™ 4mm x 33G Pen Needles
Brief Title: Comparative User Experiences With BD Nano™ PRO 4mm x 32G Extra Thin Wall Pen Needle vs Three Commercially Available Pen Needles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DBC-18PENDL02
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Results first posted 2020-03-09 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-02

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: BD Nano (Test Device) will be compared to other currently marketed devices (controls) through a series of abdominal saline injections
Who Masked: Participant
Masking Description: Participants will not see any labeling for the Pen Needles used for the injections
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- BD Nano™ PRO pen needle vs 33G Artsana Insupen Extr3me (Experimental): Subjects are to perform 2 pairs of injections. Each Pair consists of BD Nano™ PRO pen needle vs Artsana Insupen Extr3me 4mm x 33G x 2
  Interventions: Device: BD Nano™ PRO; Device: 33G Artsana Insupen Extr3me
- BD Nano™ PRO pen needle vs 34G Artsana Insupen Extr3me (Experimental): Subjects are to perform 2 pairs of injections. Each pair consists of Nano™ PRO pen needle vs Artsana Insupen Extr3me 3.5mm x 34G x 2
  Interventions: Device: BD Nano™ PRO; Device: 34G Artsana Insupen Extr3me
- BD Nano™ PRO pen needle vs Simple Diagnostics Comfort EZ™ (Experimental): Subjects are to perform 2 pairs of injections. Each pair consists of BD Nano™ PRO pen needle vs Simple Diagnostics Comfort EZ™ 4mm x 33G x 2
  Interventions: Device: BD Nano™ PRO; Device: Simple Diagnostics Comfort EZ™

INTERVENTIONS:
Device: BD Nano™ PRO — Insulin Pen needle
Device: 33G Artsana Insupen Extr3me — Insulin Pen Needle
  Arms: BD Nano™ PRO pen needle vs 33G Artsana Insupen Extr3me
Device: 34G Artsana Insupen Extr3me — Insulin Pen Needle
  Arms: BD Nano™ PRO pen needle vs 34G Artsana Insupen Extr3me
Device: Simple Diagnostics Comfort EZ™ — Insulin Pen Needle
  Arms: BD Nano™ PRO pen needle vs Simple Diagnostics Comfort EZ™

SUMMARY:
This is a subject partially blinded, block randomized, prospective, single-visit, multi-center study to compare user experiences with BD Nano™ PRO pen needle vs. three (3) thinner commercially available comparator pen needles (Artsana Insupen Extr3me 33G, Artsana Insupen Extr3me 34G and the Simple Diagnostics Comfort EZ™ 33G Pen Needles). The study will include up to 146 study subjects having Type 1 or Type 2 diabetes.

DETAILED DESCRIPTION:
The study will consist of one 60 to 120 minute visit in which pre-set doses of saline will be abdominally delivered by Subjects via a reusable insulin pen device. All pen needles will be attached by study staff. The pen needle outer cover and inner shield will be removed prior to subject use so that they will not be able to identify which device they are using. Subjects are to perform 12 injections into the abdomen (6 pairs of injections). Pairs of injections will be evaluated and each pair will contain one BD Nano™ PRO and one comparator pen needle. Within the 12 injections, each comparator will be injected twice, therefore each subject will experience 2 of each of the following pairs:

BD Nano™ PRO pen needle vs Artsana Insupen Extr3me 4mm x 33G x 2 BD Nano™ PRO pen needle vs Artsana Insupen Extr3me 3.5mm x 34G x 2 BD Nano™ PRO pen needle vs Simple Diagnostics Comfort EZ™ 4mm x 33G Each Subject will evaluate pain after completion of each pair of injections using a 15 cm relative Visual Analog Scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 75 years of age (inclusive)
2. Diagnosed with Type 1 or Type 2 diabetes
3. Self-injecting using an injection pen for ≥3 months with any pen needle
4. Injecting a minimum of ≥10 units of insulin and/or Victoza at least once per day
5. Able to demonstrate proficiency using an injection pen into an injection model
6. Able and willing to provide informed consent
7. Able and willing to complete all study procedures

Exclusion Criteria:

* a. Not self-injecting (example, injections completed by a family member) b. Self-injecting with a pen injector for less than 3 months c. Unwilling to inject into abdomen d. Unwilling to have hair at the injection area reduced with an electric razor if it is determined the hair will interfere with leakage evaluation e. Failure to confirm which pen needle (gauge and needle length) subject is currently using. To confirm, subject may be asked to bring their pen and pen needles to the site or site staff may confirm via medical record or pharmacy.

  f. Pregnant (self-attestation) g. Currently taking anti-platelet or anticoagulant therapy (up to 162 mg per day of aspirin is permitted).

  h. History of a bleeding disorder i. History of recurrent dermatological conditions or skin disorder (e.g., psoriasis, eczema) j. Gross skin anomalies and abnormalities located at or very close to the injection sites that would significantly limit available injection space.

  k. History of symptomatic low blood pressure or history of fainting (syncope) during hypodermic injections l. Use of any analgesic medications (prescription or OTC) within 24 hours of first study injection, and during the study (up to 162 mg per day of aspirin is permitted).

  m. A current or previous medical or physical condition that, in the opinion of the investigator, would place the patient at risk or make them unable to perform study procedures or has the potential to confound interpretation of the study results n. Currently participating in another pen needle study o. Employed by, or currently serving as a contractor or consultant to BD or any diabetes injectable medication, injection pen, or pen needle manufacturer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - East West Medical Research Institute, Honolulu, Hawaii
  - TKL Research Inc., Fair Lawn, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gibney MA, Fitz-Patrick D, Klonoff DC, Whooley S, Lu B, Yue W, Glezer S. User experiences with second-generation 32-gauge x 4 mm vs. thinner comparator pen needles: prospective randomized trial. Curr Med Res Opin. 2020 Oct;36(10):1591-1600. doi: 10.1080/03007995.2020.1803248. Epub 2020 Aug 18. PMID 32723109

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each subject received more than one treatment
Groups:
- All Study Participants: Subjects are to perform 6 pairs of injections. Each Pair consists of BD Nano™ PRO pen needle vs Artsana Insupen Extr3me 4mm x 33G or Artsana Insupen Extr3me 3.5mm x 34G or Simple Diagnostics Comfort EZ™ 4mm x 33G
Period: Overall Study
Arm/Group | All Study Participants
Started | 158
Completed | 154
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Protocol defined | 2
Not completed — Improper consent documentation | 1

BASELINE CHARACTERISTICS:
Population: the subject that withdrew was not counted in population because the subject withdrew before enrollment
Arm/Group | All Study Participants
Number analyzed (Participants) | 157
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 80
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 145
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 12
  Black or African American | 16
  White | 88
  More than one race | 16
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Injection Site Pain for BD Nano PRO Needle Compared to Each of Three (3) Commercially Available Comparators
Description: Injection pain as measured by a relative visual analog scale. This endpoint analyzes data for individual groups. User preference is assessed through a single question reported on a 150mm relative VAS scale with the BD Nano™ PRO pen needle Pen labeled at +75 mm and the Comparator pen needle labeled at -75mm. On this scale, zero represents no preference to either pen needle. Relative VAS scores range from -75mm to 75mm; positive scores reflect preference forBD Nano™ PRO and negative scores reflect preference for the comparator.
  Scores from each of the paired injections (308 pairs for all participants) were pooled and a mean was calculated. The two-sided 95% confidence interval was calcuated for the average relative rating. A linear model was used to adjust for the order effect.
  If the lower bound of the 95% CI is > -10cm, non-inferiority could be concluded. If the lower bound of the 95% CI is >0, superiority can also be concluded.
Time Frame: Scores were collected immediately after each paired injection
Population: Per-protocol population
Measure: Mean (95% Confidence Interval); unit: mm
Units Other Than Participants: paired injections
Arm/Group | BD Nano™ PRO Pen Needle vs 34G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs 33G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs Simple Diagnostics Comfort EZ™
Number analyzed (Participants) | 154 | 154 | 154
Number analyzed (paired injections) | 308 | 308 | 308
mm | 17.55 [11.43 to 23.67] | 17.39 [11.28 to 23.51] | 9.13 [3.01 to 15.25]

2. Secondary Outcome: Needle Bending in BD Nano™ PRO vs Each of 3 Comparator Pen Needles
Description: Participants reported a visual score of needle bending. A score of at least 2, corresponding to >10 degrees of bending, was considered an event of a bent needle. Scores from each injection (308 for each needle type) were pooled and a mean was calculated. The incidence of bent needle events in the BD Nano™ PRO and each competitor were compared and the mean difference reported with a 95% confidence interval.
Time Frame: Scores were collected immediately after each paired injection
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: Difference in incidence
Units Other Than Participants: paired injections
Arm/Group | BD Nano™ PRO Pen Needle vs 34G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs 33G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs Simple Diagnostics Comfort EZ™
Number analyzed (Participants) | 154 | 154 | 154
Number analyzed (paired injections) | 308 | 308 | 308
Difference in incidence | -0.39 [-1.82 to 1.04] | 0.13 [-2.8 to 3.06] | 0.42 [-1.91 to 2.75]
Statistical Analysis 1: Comparison: BD Nano™ PRO Pen Needle vs 34G Artsana Insupen Extr3me; Test type: Superiority — The average difference in incidence of needle bending with BD Nano vs. Comparator pen needle was calculated with 95% confidence interval and assessed for statistical significance; p = 0.591, Fisher Exact; Risk Difference (RD) = -0.39, 95% CI 2-sided [-1.82 to 1.04]
Statistical Analysis 2: Comparison: BD Nano™ PRO Pen Needle vs 33G Artsana Insupen Extr3me; Test type: Superiority — The average difference in percentage of occurrence with BD Nano vs. Comparator pen needle was calculated with 95% confidence interval and assessed for statistical significance; p = 0.931, Fisher Exact; Risk Difference (RD) = 0.13, 95% CI 2-sided [-2.8 to 3.06]
Statistical Analysis 3: Comparison: BD Nano™ PRO Pen Needle vs Simple Diagnostics Comfort EZ™; Test type: Superiority — [test comment as in outcome 2, analysis 2]; p = 0.723, Fisher Exact; Risk Difference (RD) = 0.42, 95% CI 2-sided [-1.91 to 2.75]

3. Secondary Outcome: Superiority of BD Nano™ PRO vs Each of 3 Comparator Pen Needles (Leakage)
Description: After saline delivery equivalent to 30U of U100 insulin (0.3mL) and subject removal of pen needle from body, study staff used the provided materials and scale to absorb leakage from the pen needle tip and injection site to measure the amount of leakage. Leakage over 0.015g was counted as an event. The incidence of leakage (yes/no) was calculated for each groups and the mean difference calculated along with a 95% confidence interval. A positive score indicates fewer leakage events with the BD Nano™ PRO and a negative score indicates fewer leakage events with the competitor. Scores from each injection (308 for each needle type) were pooled and a mean was calculated. The incidence of needle leakage in the BD Nano™ PRO and each comparator were compared and the mean difference reported with a 95% confidence interval.
Time Frame: Leakage was measured directly after each injection
Population: Per protocol population
Measure: Number (95% Confidence Interval); unit: Difference in incidence
Units Other Than Participants: Pen Needles
Arm/Group | BD Nano™ PRO Pen Needle vs 33G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs 34G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs Simple Diagnostics Comfort EZ™
Number analyzed (Participants) | 154 | 154 | 154
Number analyzed (Pen Needles) | 308 | 308 | 308
Difference in incidence | -5.70 [-9.0 to -3.5] | -14.09 [-26.49 to -1.69] | -0.20 [-1.9 to 0.6]
Statistical Analysis 1: Comparison: BD Nano™ PRO Pen Needle vs 33G Artsana Insupen Extr3me; Test type: Superiority — The average difference in percentage of occurrence with BD Nano vs. comparator was calculated with 95% confidence interval and assessed for statistical significance; p < 0.001, Fisher Exact; Risk Difference (RD) = -5.70, 95% CI 2-sided [-9.0 to -3.5]
Statistical Analysis 2: Comparison: BD Nano™ PRO Pen Needle vs 34G Artsana Insupen Extr3me; Test type: Superiority — [test comment as in outcome 3, analysis 1]; p = 0.026, Fisher Exact — Although a site difference was detected - all sites combined p-value was generated,; Risk Difference (RD) = -14.09, 95% CI 2-sided [-26.49 to -1.69]
Statistical Analysis 3: Comparison: BD Nano™ PRO Pen Needle vs Simple Diagnostics Comfort EZ™; Test type: Superiority — The average difference in percentage of occurrence with BD Nano vs.Comparator pen needle was calculated with 95% confidence interval and assessed for statistical significance; p = 0.644, Fisher Exact; Risk Difference (RD) = -0.20, 95% CI 2-sided [-1.9 to 0.6]

4. Secondary Outcome: Compare BD Nano™ PRO vs Each of 3 Comparator Pen Needles (Force)
Description: Subject perceived force required to deliver dose; measured by a relative 5 point Likert scale. The scale ranged from -2 to 2, where positive scores indicated less thumb force required for the BD Nano™ PRO, and negative scores indicated less thumb force for the comparator. Scores from each of the paired injections were pooled and a mean was calculated.
Time Frame: Immediately after injection Pair
Population: Subjects protocol population with non-missing data
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Units Other Than Participants: paired injections
Arm/Group | BD Nano™ PRO Pen Needle vs 33G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs 34G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs Simple Diagnostics Comfort EZ™
Number analyzed (Participants) | 154 | 154 | 154
Number analyzed (paired injections) | 306 | 305 | 307
Score on a scale | 0.8 [0.62 to 0.98] | 1.0 [0.8 to 1.16] | 0.3 [0.13 to 0.49]
Statistical Analysis 1: Comparison: BD Nano™ PRO Pen Needle vs 33G Artsana Insupen Extr3me; Test type: Superiority — Two-sided 95% confidence intervals is calculated for the average relative rating. A linear model was used to evaluate the pen needle group effect on the response to test whether the groups can be combined (a p-value < 0.05 for the pen needle group effect indicates non-poolability) and to adjust for the order effect. The order of the pen needles used and the group to which the subject belongs were used as covariates; Overall Mean = 0.8, 95% CI 2-sided [0.62 to 0.98]
Statistical Analysis 2: Comparison: BD Nano™ PRO Pen Needle vs 34G Artsana Insupen Extr3me; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Overall Mean = 1.0, 95% CI 2-sided [0.8 to 1.16]
Statistical Analysis 3: Comparison: BD Nano™ PRO Pen Needle vs Simple Diagnostics Comfort EZ™; Test type: Superiority — [test comment as in outcome 4, analysis 1]; Overall Mean = 0.3, 95% CI 2-sided [0.13 to 0.49]

5. Other Pre Specified Outcome: Compare BD Nano™ PRO vs Each of 3 Comparator Pen Needles (Total Injection Time)
Description: Time from when subject when is depressed and time when removed from body.
Time Frame: Time of injection
Population: Per Protocol Population
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Pen needles
Groups:
- All Study Participants: Subjects are to perform 6 pairs if injections. Each Pair consists of BD Nano and one comparator. Each comparator was used twice
Arm/Group | All Study Participants
Number analyzed (Participants) | 154
Number analyzed (Pen needles) | 1848
seconds
  BD NANO | 8.39 (5.26)
  Artsana 33G | 10.98 (2.64)
  Arstana 34G | 9.93 (5.16)
  Comfort EZ 33G | 8.63 (5.30)
Statistical Analysis 1: Comparison: All Study Participants; BD Nano Pro vs Artsana 34G; Test type: Superiority — A mixed effect model was used (fixed effects of PN, abdomen site, order of pair, order of PN within pair and random subject effect) to estimate average difference (BD Nano PN - Comparator PN) in delivery time and total injection time. A Box-Cox transformation might be used to normalize the data if necessary; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.192, 95% CI 1-sided [upper limit -0.141]
Statistical Analysis 2: Comparison: All Study Participants; BD NANO vs Artsana 33G. A significant site effect was detected at one site; the most conservative p-value is reported; Test type: Superiority — [test comment as in outcome 5, analysis 1]; p = 0.104, Mixed Models Analysis; Mean Difference (Final Values) = -0.122, 95% CI 1-sided [upper limit 0.016]
Statistical Analysis 3: Comparison: All Study Participants; BD NANO vs Comfort EZ 33G; Test type: Superiority — A mixed effect model was used (fixed effects of PN, abdomen site, order of pair, order of PN within pair and random subject effect) to estimate average difference (BD Nano PN - Comparator PN) in delivery time and total injection time. A Box-Cox transformation might be used to normalize the data if necessary. The upper bound of the confidence interval was compared to 0; p = 0.003, Mixed Models Analysis; Mean Difference (Net) = -0.068, 95% CI 1-sided [upper limit -0.017]

6. Post Hoc Outcome: Compare BD Nano™ PRO vs Each of 3 Comparator Pen Needles (Needle Breaking)
Description: A needle was considered broken if the patient end and canula was separated into 2 pieces. The number and proportion of needle breaking occurrence for each pen needle type were summarized. The incidence of broken needle events for the BD Nano PRO was compared to each of the 3 comparator products and the mean difference reported with a 95% confidence interval.
Time Frame: Immediately after injection
Population: Per Protocol Population
Measure: Mean (95% Confidence Interval); unit: Difference in incidence
Units Other Than Participants: paired injections
Arm/Group | BD Nano™ PRO Pen Needle vs 33G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs 34G Artsana Insupen Extr3me | BD Nano™ PRO Pen Needle vs Simple Diagnostics Comfort EZ™
Number analyzed (Participants) | 154 | 154 | 154
Number analyzed (paired injections) | 308 | 308 | 308
Difference in incidence | 0 [-0.4 to 1.2] | 0 [-0.4 to 1.2] | 0 [-0.4 to 1.2]
Statistical Analysis 1: Comparison: BD Nano™ PRO Pen Needle vs 33G Artsana Insupen Extr3me; Test type: Superiority — The number and proportion of needle breaking occurrence for each pen needle type were summarized. A 95% confidence interval for difference in proportions between BD Nano Pro and the Comparator was calculated using the score method for independent proportions; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.4 to 1.2]
Statistical Analysis 2: Comparison: BD Nano™ PRO Pen Needle vs 34G Artsana Insupen Extr3me; Test type: Superiority — [test comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.4 to 1.2]
Statistical Analysis 3: Comparison: BD Nano™ PRO Pen Needle vs Simple Diagnostics Comfort EZ™; Test type: Superiority — [test comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.4 to 1.2]

7. Post Hoc Outcome: Subject Satisfaction Survey
Description: Each subject was given a non-comparative 4-question survey on Pen needle characteristics.
Time Frame: At the end of study
Population: Each subject was provided a 4 question survey of their general experience with pen needles. The questions were based on a a 5 point type of Likert scale.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 154
Participants
  Injection pain affects my level of satisfaction: Agree | 56
  Injection pain affects my level of satisfaction: Somewhat Agree | 46
  Injection pain affects my level of satisfaction: Neutral | 27
  Injection pain affects my level of satisfaction: Somewhat disagree | 8
  Injection pain affects my level of satisfaction: Disagree | 17
  Thumb pressure affects my level of satisfaction: Agree | 54
  Thumb pressure affects my level of satisfaction: Somewhat Agree | 51
  Thumb pressure affects my level of satisfaction: Neutral | 26
  Thumb pressure affects my level of satisfaction: Somewhat disagree | 9
  Thumb pressure affects my level of satisfaction: Disagree | 14
  Post injection leakage affects my level of concern: Agree | 76
  Post injection leakage affects my level of concern: Somewhat Agree | 31
  Post injection leakage affects my level of concern: Neutral | 23
  Post injection leakage affects my level of concern: Somewhat disagree | 8
  Post injection leakage affects my level of concern: Disagree | 16
  A bend needle increases my level of concern: Agree | 100
  A bend needle increases my level of concern: Somewhat Agree | 28
  A bend needle increases my level of concern: Neutral | 13
  A bend needle increases my level of concern: Somewhat disagree | 2
  A bend needle increases my level of concern: Disagree | 11

ADVERSE EVENTS:
Time Frame: one day
Groups:
- BD Nano™ PRO Pen Needle; 34G Artsana Insupen Extr3me; 33G Artsana Insupen Extr3me; Simple Diagnostics Comfort EZ™: Subjects are to perform 2 pairs of injections. Each pair consists of Nano™ PRO pen needle vs a competitor product.
Arm/Group | BD Nano™ PRO Pen Needle | 34G Artsana Insupen Extr3me | 33G Artsana Insupen Extr3me | Simple Diagnostics Comfort EZ™
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/157 | 0/157 | 0/157
Serious Adverse Events (participants affected / at risk) | 0/157 | 0/157 | 0/157 | 0/157
Other Adverse Events (participants affected / at risk) | 0/157 | 0/157 | 0/157 | 0/157

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT03878758/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-30): https://cdn.clinicaltrials.gov/large-docs/58/NCT03878758/SAP_001.pdf